CLINICAL TRIAL: NCT05874895
Title: MAnual Lymphatic DrAinage to iMprove the outcomE of Patients After Septic Shock: A Safety and Feasibility Pilot Randomized Controlled Trial
Brief Title: MAnual Lymphatic DrAinage to iMprove the outcomE of Patients After Septic Shock
Acronym: MADAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MADAME trial
Record Dates: First submitted 2023-05-11; First posted 2023-05-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Multiorgan Failure; Inflammatory Response; Septic Shock
Keywords: Sepsis; Multiorgan Failure; Excessive Inflammatory Response; Manual Lymphatic Drainage; Lymphatic System; Septic Shock
MeSH Terms: conditions — Sepsis; Multiple Organ Failure; Shock, Septic | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: The study subjects will be randomized in two study arms.
Masking Description: No masking will be used in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Lymphatic Drainage (Experimental): In addition to usual care, daily manual lymphatic drainage will be performed for five consecutive days. After this period.
  Interventions: Procedure: Manual Lymphatic Drainage
- Usual Care (Active Comparator): Usual care for patients with septic shock will be provided.
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: Manual Lymphatic Drainage — Manual lymphatic drainage massage involves gently manipulating specific areas of the body to help lymph move to an area with working lymph vessels.
  Arms: Manual Lymphatic Drainage
Procedure: Usual Care — Usual care provided for patients in septic shock.
  Arms: Usual Care

SUMMARY:
Antimicrobial and supportive therapeutic interventions in patients with septic shock are usually effective - procalcitonin and interleukin-6 levels fall rapidly in most cases, and noradrenaline support can be discontinued within a few days. Unfortunately, only in a small portion of patients, do the organ functions improve at the same time, and in most of them, multi-organ failure persists. Therefore, it is likely that, in addition to infection and the response to infection, other mechanisms are also involved in the persistence of organ failure in patients after septic shock.

DETAILED DESCRIPTION:
One of the possible explanations for prolonged multi-organ dysfunction after an excessive inflammatory phase is a disorder of "post-inflammatory cleaning", the so-called resolution of inflammation. The resolution of inflammation is a regulated process in which the controlling action of specialized pro-resolution mediators (lipoxins, resolvins, etc.), conversion of pro-inflammatory macrophages (M1) to pro-resolution (M2., induce the process of structural tissue restoration), autophagy plays a significant role and, of course, the flushing of accumulated interstitial fluid with waste products by lymphatic drainage. Any disturbance in pro-resolution mechanisms can lead to prolonged organ dysfunction.

The lymphatic system plays a key role in maintaining fluid homeostasis. Its ability to drain interstitial fluid can increase up to 20 times. However, even such an increase may not be sufficient in the situation of extreme interstitial fluid sequestration that accompanies septic shock. In addition, some inflammatory mediators (for example, nitric oxide, TNF-α, Interleukin-1β) cause relaxation of the vascular structures of the lymphatic system, slowing the flow of lymph. The result is the persistence of tissue swelling with tissue hypoxia due to the extension of the diffusion path for oxygen and the accumulation of waste products of inflammation.

Manual lymphatic drainage (MLD) is one of the treatments that stimulate the lymphatic system. In general, it is expected to accelerate the outflow of lymph and waste products from tissues previously affected by inflammation, accelerate the recovery of tissue function, sympatholytic effect and increase the tension of the vagus nerve. It can therefore be assumed that MLD will have a beneficial effect on the course of persistent multi-organ dysfunction in patients after therapeutically managed septic shock.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of septic shock at admission to ICU
* sepsis or suspicion of sepsis
* noradrenaline support required in order to maintain mean arterial pressure ≥ 65 mmHg
* serum lactate ≥ 2 mmol/L

Exclusion Criteria:

* patients <18 years of age
* pregnant women with septic shock, in whom the pregnancy has been preserved
* patients with a history of heart failure with NYHA (New York Heart Association) classification ≥ III
* patients with a history of thromboembolic events
* patients with septic shock transferred from another department/hospital, if the length of stay at the previous workplace exceeded 72 hours
* patients with septic shock and an inauspicious prognosis, or in the phase of withdrawal of treatment
* patients with uncontrolled infection
* patients with septic shock who lack informed consent
* patients with septic shock, in whom the SOFA score decreased by more than 50% during the day following the withdrawal of noradrenaline (i.e. a subgroup of patients with a rapid improvement of the clinical course after the resolution of septic shock).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Feasibility Outcome - number of patients undergoing manual lymphatic drainage procedure. | 12 months
  The anticipated number of patients is 2 per month.
Feasibility Outcome - The percentage of patients suitable for manual lymphatic drainage procedure in whom this procedure has been performed. | 12 months
  It is expected that manual lymphatic drainage procedure will be performed in at least 80 per cent of patients.
Safety Outcome - the percentage of cases when the manual lymphatic drainage procedure interferes with standard nursing care | 12 months
  interference is assumed in 0 per cent of cases
Safety Outcome - incidence of the need to restart circulatory support with norepinephrine | 12 months
  The presumed incidence is assumed in 0 per cent of cases
Safety Outcome - incidence of thromboembolic events | 12 months
  The presumed incidence is assumed in 0 per cent of cases
Efficacy Outcome - change in SOFA (sequential organ failure assessment) score | 12 months
  Comparison of the SOFA score on Days 3 and 5 versus Day 0 (randomisation day)
Efficacy Outcome - incidence of delirium | 12 months
  Incidence of delirium for the period from randomisation until discharge from ICU
Efficacy Outcome - 28-day mortality | 12 months
  28-day mortality will be observed

CONTACTS AND LOCATIONS:
Overall Officials: Roman Kula, MD,CSc, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Alitalo K. The lymphatic vasculature in disease. Nat Med. 2011 Nov 7;17(11):1371-80. doi: 10.1038/nm.2545. PMID 22064427
- [Background] Venero Galanternik M, Stratman AN, Jung HM, Butler MG, Weinstein BM. Building the drains: the lymphatic vasculature in health and disease. Wiley Interdiscip Rev Dev Biol. 2016 Nov;5(6):689-710. doi: 10.1002/wdev.246. Epub 2016 Aug 30. PMID 27576003
- [Background] Oliver G, Kipnis J, Randolph GJ, Harvey NL. The Lymphatic Vasculature in the 21st Century: Novel Functional Roles in Homeostasis and Disease. Cell. 2020 Jul 23;182(2):270-296. doi: 10.1016/j.cell.2020.06.039. PMID 32707093
- [Background] Vairo GL, Miller SJ, McBrier NM, Buckley WE. Systematic review of efficacy for manual lymphatic drainage techniques in sports medicine and rehabilitation: an evidence-based practice approach. J Man Manip Ther. 2009;17(3):e80-9. doi: 10.1179/jmt.2009.17.3.80E. PMID 20046617
- [Background] Scallan JP, Zawieja SD, Castorena-Gonzalez JA, Davis MJ. Lymphatic pumping: mechanics, mechanisms and malfunction. J Physiol. 2016 Oct 15;594(20):5749-5768. doi: 10.1113/JP272088. Epub 2016 Aug 2. PMID 27219461
- [Background] Klaourakis K, Vieira JM, Riley PR. The evolving cardiac lymphatic vasculature in development, repair and regeneration. Nat Rev Cardiol. 2021 May;18(5):368-379. doi: 10.1038/s41569-020-00489-x. Epub 2021 Jan 18. PMID 33462421
- [Background] Pruitt LG. Lymphatic flow modulation as adjunct therapy for septic shock. Med Hypotheses. 2020 Sep;142:109748. doi: 10.1016/j.mehy.2020.109748. Epub 2020 Apr 20. PMID 32339860
- [Background] Vieira JM, Norman S, Villa Del Campo C, Cahill TJ, Barnette DN, Gunadasa-Rohling M, Johnson LA, Greaves DR, Carr CA, Jackson DG, Riley PR. The cardiac lymphatic system stimulates resolution of inflammation following myocardial infarction. J Clin Invest. 2018 Aug 1;128(8):3402-3412. doi: 10.1172/JCI97192. Epub 2018 Jul 9. PMID 29985167
- [Background] Frohlich E. Acute Respiratory Distress Syndrome: Focus on Viral Origin and Role of Pulmonary Lymphatics. Biomedicines. 2021 Nov 20;9(11):1732. doi: 10.3390/biomedicines9111732. PMID 34829961
- [Background] Schwager S, Detmar M. Inflammation and Lymphatic Function. Front Immunol. 2019 Feb 26;10:308. doi: 10.3389/fimmu.2019.00308. eCollection 2019. PMID 30863410
- [Background] Kraft JD, Blomgran R, Lundgaard I, Quiding-Jarbrink M, Bromberg JS, Borgeson E. Specialized Pro-Resolving Mediators and the Lymphatic System. Int J Mol Sci. 2021 Mar 9;22(5):2750. doi: 10.3390/ijms22052750. PMID 33803130
- [Background] Fanous MY, Phillips AJ, Windsor JA. Mesenteric lymph: the bridge to future management of critical illness. JOP. 2007 Jul 9;8(4):374-99. PMID 17625290
- [Background] Wu C, Li H, Zhang P, Tian C, Luo J, Zhang W, Bhandari S, Jin S, Hao Y. Lymphatic Flow: A Potential Target in Sepsis-Associated Acute Lung Injury. J Inflamm Res. 2020 Nov 23;13:961-968. doi: 10.2147/JIR.S284090. eCollection 2020. PMID 33262632